CLINICAL TRIAL: NCT07162389
Title: Early Stability of Short Dental Implants With Shallow Threads in the Posterior Mandible: A Controlled Clinical Pilot Study .
Brief Title: Comparative (Short vs. Standard) Length Implants in Early Stability Patterns.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Science and Technology, Yemen (Other)
Responsible Party: Principal Investigator, Mohammad A Al-Jonaid M.Sc., M.Sc Candidate in Oral Surgery and implantology, University of Science and Technology, Yemen
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1447/0062/UREC/UST.
Record Dates: First submitted 2025-07-18; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Alveolar Bone Atrophy
Keywords: RFA; ISQ; Short dental implants; Shallow-threaded; Posterior Mandible; Early Dynamic Changes; primary Stability; Stability dip
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: Interventional Study A Prospective, controlled, parallel-group, anatomically allocated pilot study
  . Anatomically-Driven Allocation
  * Group A (Short Implants): 7mm implants placed in sites with 8.5-9mm residual bone height (measured from crest to inferior alveolar nerve + 1.5mm safety margin).
  * Group B (Standard Implants): 11mm implants placed in sites with ≥12.5mm bone height.
  * Rationale: Mimics real-world clinical decision-making where implant length is determined by available bone anatomy.
    2. Technical Controls:
  * Standardized diameter: All implants 4.2mm (Tiologic Twinfit system).
  * Identical surface/macrodesign: SLA surface, shallow threads (<0.5mm depth), reverse-buttress profile.
  * Surgical calibration: Single operator, under-drilling protocol for D2 bone (final drill -0.2mm), non-condensing drilling for D3 bone.
    3. Dynamic Monitoring Protocol:
  * Timepoints: T0 immediate, T1,T2,T3,T4 (at the end of weeks- 1,2,3,4)
Who Masked: Outcomes Assessor
Masking Description: This clinical trial employs partial masking (blinding) to minimize bias in outcome assessments:
  1. Blinded Parties
     * Outcome Assessors:
     * The researcher performing resonance frequency analysis (RFA) measurements (ISQ values at T0-T4) is masked to:
     * Implant length (7mm vs. 11mm)
     * Insertion torque value (ITV) Rationale: Prevents measurement bias in stability tracking.
     * Data Analysts:
     * Statisticians processing ISQ trends are blinded to group allocation until analysis completion.
  2. Non-Blinded Parties
     * Surgeon: Cannot be masked due to visual/tactile differences during osteotomy preparation.
     * Patients: Aware of implant type due to post-operative healing abutment visibility.
  3. Blinding Methods
     * RFA Protocol:
     * SmartPeg placement/readings performed by a separate researcher not involved in surgery.
     * ISQ values recorded using coded forms without implant length details.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Short Dental Implant Group. (Experimental): Group A, Shallow-Threaded ,length 7mm, diameter 4.2mm,10 single dental implants.
  Interventions: Device: Shallow-Threaded Short Implant (SHI); Device: Shallow-Threaded Standard Implant (SDI)
- Standard Dental Implant Group. (Active Comparator): Group B, Shallow-Threaded ,length 11mm, diameter 4.2mm,10 single dental implants.
  Interventions: Device: Shallow-Threaded Short Implant (SHI); Device: Shallow-Threaded Standard Implant (SDI)

INTERVENTIONS:
Device: Shallow-Threaded Short Implant (SHI) — A 7mm long, 4.2mm diameter dental implant with shallow thread (<0.5mm depth) Macrodesign, surgically placed in the jawbone to restore missing teeth
Device: Shallow-Threaded Standard Implant (SDI) — A 11mm long, 4.2mm diameter dental implant with shallow thread (<0.5mm depth) macrodesign, surgically placed in the jawbone to restore missing teeth.

SUMMARY:
Early Stability of Short vs. Standard Dental Implants in the Posterior Mandible

This study compares how well short dental implants (7mm) work compared to standard-length implants (11mm) when placed in the back part of the lower jaw. Both types of implants have special shallow threads designed to reduce stress on the bone. The main goal is to see how stable they are during the first 4 weeks after placement-a critical time for healing.

* Short implants may be a good option for patients with limited jawbone height, avoiding the need for bone grafting.
* Understanding their early stability helps dentists decide when it's safe to place teeth on them.
* This study uses advanced tools like 3D scans (CBCT) and implant stability measurements (ISQ) to track healing.

What will happen in the study?

1. Screening: A dental exam and 3D scan to check bone quality.
2. Implant Placement:

   * Short (7mm) or standard (11mm) implant, depending on your bone height.
   * Minimally invasive surgery with local anesthesia.
3. Follow-ups: Painless stability checks at end of 1, 2, 3, and 4 weeks using a small device (RFA).

Who can participate?

Adults (18-60 years) missing posterior teeth in the lower jaw, with:

* Enough bone width (≥6.5mm).
* No uncontrolled health conditions (e.g., severe diabetes).
* Non-smokers or light smokers (<10 cigarettes/day).
* Benefits: Free implant placement and monitoring; contributes to better dental care.
* Risks: Typical surgery risks (swelling, infection); rare nerve injury (<5% chance).

How long is the study?

* Active participation: 4 weeks (with optional long-term follow-up).
* Total study duration: ~12 months (including data analysis). Mohammad Abdulwahab Al-Jonaid University of Science and Technology, Sana'a.
* Supervisor: Dr. Ali Al-Hudaied, Oral and Maxillofacial Surgery Specialist.

DETAILED DESCRIPTION:
A prospective, controlled, parallel-group pilot clinical trial comparing 7mm short implants (SHI) versus 11mm standard implants (SDI) with identical shallow-thread macrodesign (depth <0.5mm) and 4.2mm diameter. Implant allocation is anatomically driven based on CBCT-measured vertical bone height (7mm group: 8.5-9mm residual bone; 11mm group: ≥12.5mm).

Technical Innovations

1. Thread Geometry: Dual shallow-thread reverse-buttress design (0.2-0.5mm depth) with progressive pitch to optimize cortical engagement while minimizing shear stress (Ao et al. 2010).
2. Surgical Protocol: Standardized osteotomy using under-drilling for D2 bone (final drill diameter reduced by 0.2mm) and non-condensing drilling for D3 bone to prevent over-compression.
3. Stability Metrics:

   * Primary Stability: ITV (last quarter-turn torque) + ISQ (Penguin RFA, mean of 4-directional measurements).
   * Dynamic Stability: ISQ tracked at T0 (baseline), T1 (7d), T2 (14d), T3 (21d), T4 (28d) to capture dip magnitude (ΔISQ) and recovery onset (start of biological stability).

Bone Density Integration

* Pre-op CBCT: Hounsfield Unit (HU) stratification (D2: 800-1250 HU; D3: 350-850 HU) with 2mm² ROI analysis at coronal/middle/apical levels.
* Intra-op Validation: Tactile assessment using Lekholm & Zarb scale (D2: "white pine" resistance; D3: "balsa wood").

Quality Controls

* Operator Standardization: Single experienced surgeon performs all placements.
* RFA Calibration: Pre-measurement checks with reference block and standardized SmartPeg torque (5-10 Ncm).
* Blinding: ISQ measurements by research assistant masked to implant type.

Rationale for 4-Week Endpoint

Focuses on the critical early healing phase where:

1. Primary stability (mechanical) transitions to secondary stability (biological).
2. The "stability dip" (week 2-4) predicts osseointegration failure risk.

Technical Constraints

* Limited Sample Size (n=20): Pilot study design prioritizes feasibility over powered comparisons.
* Bone Density Homogeneity: Excludes D1/D4 bone to reduce confounding.

Innovative Aspects

First clinical study to combine:

1. Shallow threads + short length in posterior mandible.
2. Weekly RFA tracking during the dip phase.
3. HU-quantified bone density correlation with ISQ trends.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults ≥18 years with partial posterior mandibular edentulism. 2. Bone height ≥7 mm and width >6 mm (CBCT-confirmed). 3. D2/D3 bone density (HU: 350-1250). 4. Healed posterior mandibular sites (3-6 months post-extraction). 5. Good oral hygiene (plaque index ≤1). 6. Willingness to adhere to study protocols.

Exclusion Criteria:

* 1. Uncontrolled systemic diseases (e.g., diabetes with HbA1c >7%, liver disease) or medications affecting bone healing (e.g., corticosteroids, bisphosphonates).

  2. History of head/neck radiotherapy (with in past year). 3. Heavy smoking (>10 cigarettes/day). 4. Absolute contraindications for oral surgery (e.g., recent MI/CVA < 6months, bleeding disorders).

  5. Active periodontal disease, parafunctional habits as bruxism, or prior bone grafting at the site.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Implant Stability Quotient (ISQ) at Baseline (T0) | Measurement at implant placement(Day 0)
  Mean Resonance frequency Analysis(RFA) measurement taken immediately post-implantation(T0), to assess primary mechanical stability. ISQ range 1-100, low stability <60, medium stability 60 to 69, high more than or equal 70. Reported as mean ISQ value per group.
Insertion Torque value- ITV. | Measurement at during implant placement (intraoperative)
  The rotational torque in Ncm,applied during the final quarter-turn of implant insertion. This is direct measure of primary mechanical stability. Reported as mean ITV per group.
Magnitude of Stability Dip | from implant placement (Day 0) through week4
  The mean lowest point of stability curve , calculated as the greatest negative change in ISQ value from the baseline T0, measurement for each implant during the 4 -week monitoring period.
Time of Onset of Secondary Stability | from Day0 , through week 4.
  The mean time in days post implantation at which the ISQ value begins to consistently increase, indicating the start biological secondary stability. Defined as the time point after the nadir -T2or T3.where the ISQ value shows a positive increase confirmed at the subsequent measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- university of Sciences and Technology, Sanaa, Yemen

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data available upon request after publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months from 21/07/2025
Access Criteria: De-identified individual participant data will be made available upon reasonable request to corresponding author . Requests require a methodology sound proposal and a signed data access agreement.

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2025-08-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT07162389/Prot_ICF_000.pdf